CLINICAL TRIAL: NCT00364403
Title: Glycemic Load and Infant Birth Weight in Pregnant Overweight/Obese Women
Brief Title: A Low Glycemic Load Diet During Pregnancy in Overweight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Thrasher Research Fund (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: David Ludwig, MD, PhD, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R03DK073335 (NIH); R03DK073335 (NIH)
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Overweight; Pregnancy
Keywords: Glycemic index; Glycemic load; Low fat; Impaired glucose tolerance; Large for gestational age infant; Excessive body weight
MeSH Terms: conditions — Overweight; Glucose Intolerance | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Low glycemic load diet
  Interventions: Behavioral: Low glycemic load
- 2 (Active Comparator): Low fat diet
  Interventions: Behavioral: Low fat diet

INTERVENTIONS:
Behavioral: Low glycemic load — Provision of foods and dietary counseling to promote a low glycemic load diet
  Arms: 1
Behavioral: Low fat diet — Provision of foods and dietary counseling to promote a low fat diet
  Arms: 2

SUMMARY:
This study will compare the effects of a low glycemic load versus standard diet for pregnancy on outcomes related to risk for obesity, diabetes, and heart disease in both mother and infant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with prepregnant or first trimester BMI equal to or greater than 25 kg/m2 and less than 45 kg/m2
* Singleton pregnancy
* Willing to consume the diets for duration of pregnancy
* Participant to be at week 28 or less of pregnancy at baseline visit

Exclusion Criteria:

* Smoking during pregnancy
* Major medical illness (e.g., diabetes mellitus, hypertension, thyroid disease)
* Patients taking prescription medication known to affect body weight
* Alcohol consumption during pregnancy
* Patients who declare their intention to deliver infants in the environment outside of Beth Israel Deaconess Medical Center, Boston
* High level of physical activity

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Birth weight as assessed by z-scores | At birth

SECONDARY OUTCOMES:
Maternal energy intake | During pregnancy
Maternal weight gain | During pregnancy
Maternal insulin resistance assessed by HOMA | During pregnancy
Maternal metabolic syndrome components | During pregnancy
Infant body composition (ponderal index, skinfold thickness) | At birth
Cord blood glucose | At birth
cord blood insulin | At birth
cord blood leptin | At birth

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Erinn Rhodes, MD, Study Director — Boston Children's Hospital
Locations (2):
- United States (2):
  - Children's Hospital Boston, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Rhodes ET, Pawlak DB, Takoudes TC, Ebbeling CB, Feldman HA, Lovesky MM, Cooke EA, Leidig MM, Ludwig DS. Effects of a low-glycemic load diet in overweight and obese pregnant women: a pilot randomized controlled trial. Am J Clin Nutr. 2010 Dec;92(6):1306-15. doi: 10.3945/ajcn.2010.30130. Epub 2010 Oct 20. PMID 20962162